CLINICAL TRIAL: NCT06852885
Title: Evaluation of a Food Access Program on Inpatient Nutrition, Recovery, Cost of Care, and Health Related Quality of Life in Selected Public Hospitals in Rwanda
Brief Title: Evaluation of a Rwanda Hospital Feeding Program on Nutrition, Recovery, Costs of Care and Health Related Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solid'Africa (Other)
Responsible Party: Principal Investigator, Stefanie Weiland, Principal Investigator, Solid'Africa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RNEC80/2024
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Nutrition
Keywords: Nutrition; hospitals, public; malnutrition; sub-Saharan Africa; food intake
MeSH Terms: conditions — Malnutrition | interventions — Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemura (Experimental): The intervention of the Solid'Africa Gemura selective feeding program will be administered as usual for study participants in the two intervention sites. Eligible hospital inpatients will receive three meals a day during their hospital stay, as prescribed by hospital nutritionists for their specific conditions and ordered from Solid'Africa. The Solid'Africa team will prepare the ordered meals in their off-site kitchen in Rusororo and deliver them daily to the hospitals where the meals will be distributed to the study participants. Meal caloric and nutritional content information is standardized except upon request. The normal meal is 575g of food consisting of 2300kCal with 300g of carbohydrates, 175g of protein, and 100g vitamins/minerals. In addition, Solid'Africa will adjust meal content per nutritionist request for specific needs like low salt/sugar, etc.
  Interventions: Other: Meals
- Control (No Intervention): This arm includes inpatients meeting the same eligibility criteria as the intervention arm. However, no intervention will be offered and these patients will experience a hospital stay as usual.

INTERVENTIONS:
Other: Meals — The intervention of the Solid'Africa Gemura selective feeding program will be administered as usual for study participants in the two intervention sites. Eligible hospital inpatients will receive three meals a day during their hospital stay, as prescribed by hospital nutritionists for their specific conditions and ordered from Solid'Africa. The Solid'Africa team will prepare the ordered meals in their off-site kitchen in Rusororo and deliver them daily to the hospitals where the meals will be distributed to the study participants. Meal caloric and nutritional content information is standardized except upon request. The normal meal is 575g of food consisting of 2300kCal with 300g of carbohydrates, 175g of protein, and 100g vitamins/minerals. In addition, Solid'Africa will adjust meal content per nutritionist request for specific needs like low salt/sugar, etc.
  Arms: Gemura

SUMMARY:
The purpose of this interventional study was to evaluate outcomes for Solid'Africa's Gemura feeding program in four selected public hospitals comparing results between patients receiving and patients not receiving the feeding program. The study measured the effects of the program on patients nutritional status, recovery during hospitalization, patient health related-quality of life, patient satisfaction, and patient costs of care. Participants were asked: (1) to eat meals provided three times a day if they were in the intervention group; (2) to participate in an intake and discharge survey; and (3) to participate in a daily food intake survey.

DETAILED DESCRIPTION:
A multi-center, quasi-experimental study using difference-in-differences controlled comparison to test the outcomes of Solid'Africa's Gemura feeding intervention in four selected public hospitals (two in intervention group and other two in control group) from urban and peri-urban areas targeting socioeconomically vulnerable inpatients. This study has a primary outcome which is nutritional status as measured by body mass index (BMI), and secondary outcomes which include recovery during hospitalization, patient health-related quality of life (HRQOL), patient satisfaction, and patient costs of care.

ELIGIBILITY:
Inclusion Criteria:

* Hospital inpatients
* Vulnerable socioeconomic status according to social worker assessment
* Most inpatient categories
* Voluntary, self-feeding ability
* Able to stand on scale, with help if needed

Exclusion Criteria:

* Hospital outpatients
* Patients not determined socioeconomically vulnerable by social worker
* Pregnant women hospitalized for delivery
* Patients undergoing special treatment for malnutrition
* Patients receiving enteral or parenteral nutrition treatment
* Patients receiving any kind of artificial feeding support
* Patients unable to stand on scale to measure weight

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 794 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Nutritional status | Baseline and final day of patient stay, on average day 5
  Nutritional status will be measured anthropometrically in terms of weight-for-height for all participants to calculate body mass index (BMI = kg/m2). Weight will be measured with a digital weight scale and height will be measured in recumbent position for patients unable to stand and in a standing position for other patients using a height board or a tape measure. Nutritional status will also be classified at baseline and at endline, with BMI < 18.5 considered underweight, 18.5-24.9 normal weight, 25.0-29.9 overweight, and 30.0+ obese.49 Underweight will be further classified as standard for adults and for children. For children, chronic malnutrition or stunting (low height for age) and acute malnutrition or wasting (low weight for height) will be defined according to the World Health Organization growth charts and classification standards.

SECONDARY OUTCOMES:
Length of Stay | Baseline and final day of patient stay, on average day 5
  LOS will be measured in days (or fractions thereof) and collected as patient record data from routine data sources, such as patient charts, by trained research assistants.
Treatment outcome | Final day of patient stay, on average day 5
  Treatment outcome will be measured with a survey tool created to assess completion and outcome of treatment and recovery during the hospitalization period from the perspective of the attending health care worker. Questions on treatment outcome will frame answers on a Likert scale. Additional qualitative questions on treatment outcome from the patients' perspective will be included on the patient discharge survey.
Costs of treatment | Final day of patient stay, on average day 5
  Costs of treatment will be measured in RWF and collected from both heath facility records of patient treatment costs as well as from patients in their discharge survey. Where precise figures are not available or recalled, such as transportation costs, estimates may be made based on available data. Costs will be measured from the patient perspective, but may also include the health service perspective to get a societal perspective.
Patient satisfaction | Final day of patient stay, on average day 5
  Patient satisfaction will be measured with a survey on discharge including one open-ended question on satisfaction and another based on the Net Promoter Score (NPS). NPS has been widely used in business and in healthcare settings, including by the UK National Health Service (NHS). The open-ended survey question with reference to the NHS's most recently updated patient survey guidance.
Health-related quality of life | Final day of patient stay, on average day 5
  Patient health-related quality of life is measured as a patient reported outcome and surveyed using the EuroQol EQ-5D-3L (5 dimension/3 level) health questionnaire. This standardized measure of health-related quality of life developed by the EuroQol Group is a simple, generic questionnaire for use in clinical and economic appraisal or population health status surveys. Respondents answer "no/some/extreme problems" to questions in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It is a point-in-time survey and was administered by trained research assistants to participants at discharge. The Kinyarwanda version is provided by EuroQol. Part 2 is a standard vertical 20 cm visual analogue scale, used in recording an individual's rating of their overall current health-related quality of life. The scale ranges from 100 ('the best imaginable health state' or 'the best health state you can imagine') to 0 ('the worst imaginable health state').

OTHER OUTCOMES:
Food intake | Daily until final day of patient stay, about every 24 hours for 5 days on average
  In addition to nutritional status, the study will measure food intake as a patient-reported intermediate outcome measure. Trained research assistants will survey enrolled patients daily to measure estimated quantity, content, and frequency of food intake as well as a comparison to food intake at home. The food intake surveys will also provide additional qualitative data that will be used for thematic analysis and interpretation of other outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Weiland, MSc MPH, Principal Investigator
Locations (4):
- Rwanda (4):
  - Centre Hopitalier Universitaire de Butare, Butare
  - Centre Hopitalier Universitaire de Kigali, Kigali
  - Masaka Hospital, Kigali
  - Nyamata Hospital, Nyamata

IPD SHARING:
Plan to Share IPD: No
IDP may be shared upon reasonable request.